CLINICAL TRIAL: NCT05365555
Title: Analgesic Effect of Blind Fascia Iliaca Compartment Block Compared to an Ultrasound-guided Femoral Nerve Block in Patients With Hip Fractures
Brief Title: Blind Fascia Iliaca Compartment Block Compared to Ultrasound-guided Femoral Nerve Block in Patients With Hip Fractures
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Daniel Wilhelms, MD, Emergency Department Head of Research, University Hospital, Linkoeping
Other Study IDs: SE2021-05967-01
Record Dates: First submitted 2022-04-27; First posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures | interventions — Anesthesia, Conduction; Ropivacaine; Anesthetics, Local

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fascia Iliaca Compartment Block (FICB): Participants with a radiologically verified hip fracture receiving a FICB using a blind technique guided by anatomical landmarks.
  Interventions: Procedure: Fascia Iliaca Compartment Block; Drug: Ropivacaine
- Femoral Nerve Block (FNB): Participants with a radiologically verified hip fracture receiving a FNB using ultrasound guidance for direct nerve visualisation.
  Interventions: Procedure: Femoral Nerve Block; Drug: Ropivacaine

INTERVENTIONS:
Procedure: Fascia Iliaca Compartment Block — Blind technique.
  Other Names: Peripheral nerve block; Regional anesthesia
  Groups: Fascia Iliaca Compartment Block (FICB)
Procedure: Femoral Nerve Block — Ultrasound guided.
  Other Names: Peripheral nerve block; Regional anesthesia
  Groups: Femoral Nerve Block (FNB)
Drug: Ropivacaine — Ropivacaine dosed according to local guidelines.
  Other Names: Local anesthetic; Naropin

SUMMARY:
The goal of this study is to compare the analgesic effect of a blind fascia iliaca compartment block to an ultrasound-guided femoral nerve block in patients that present to the emergency department with hip fractures.

DETAILED DESCRIPTION:
Hip fractures often present to the emergency department and elderly, already fragile, patients are overrepresented. The pain associated with a hip fracture can be severe and have deleterious effects on the patient. Many studies, and a Cochrane review, have shown that a peripheral nerve block provides good pain relief and has many benefits compared to traditional pain relief, such as intravenous morphine. There is less consensus regarding which kind of nerve block, and which technique, is best to use. Many studies compared different kinds of nerve blocks to traditional methods, or more recently compared different kinds of ultrasound-guided techniques to each other.

This study proposes to compare the widely used technique of a blind fascia iliaca compartment block (FICB) to an ultrasound-guided femoral nerve block (FNB) that is currently being rolled out locally as an alternative. During the implementation period of this new clinical routine, it will be possible to compare the efficacy of FICB and FNB in reducing participant-reported pain.

ELIGIBILITY:
Inclusion Criteria:

* Adult emergency department patient over 18 years of age with a radiologically verified fracture classified as hip fracture that are eligible for a peripheral nerve block according to local guidelines

Exclusion Criteria:

* Multi-system trauma
* Isolated pelvic or diaphyseal femur fracture
* Patients unable to communicate regardless of reason
* Patients with contraindications to receiving a peripheral nerve block with an amide local anaesthetic according to local guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients in the emergency department with a radiologically verified hip fracture eligible for a peripheral nerve block according to local guidelines
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Mean Change from Baseline in Pain Scores on the Numeric Rating Scale (0 to 10, where 10 is Maximum Pain) at 30 minutes after Administration of Block, at Rest and During Active Hip Flexion | Measured 30 minutes after administered nerve block.
  Change in reported pain score should be at least one whole unit on the numeric rating scale.

SECONDARY OUTCOMES:
Ratio of Failed Blocks | Through study completion, an average of 1 year
  Defined by a failure to reduce reported pain 30 minutes after administered block by at least one whole unit on the numeric rating scale
Rate of Complications | Through study completion, an average of 1 year
  Comparing the rate of any reported complication between cohorts

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Wilhelms, PhD, MD, Principal Investigator — University Hospital, Linköping
Locations (1):
- Akutmottagningen US Östergötland, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-04-26): https://cdn.clinicaltrials.gov/large-docs/55/NCT05365555/ICF_000.pdf